CLINICAL TRIAL: NCT04706195
Title: Early Accessible Person-centred Rehabilitation With the Focus on Return to Work for Patients With Chronic Pain (EAPER-P)
Brief Title: Early Accessible Person-centred Rehabilitation for Patients With Chronic Pain
Acronym: EAPER-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EAPER-P
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: Person-centred care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred care (Experimental): PCC in the form of a combined eHealth and structured telephone support combined with an eHealth support on top of usual care
  Interventions: Behavioral: Person-centred care at distance through an eHealth platform
- Usual care (No Intervention): Regular evidence-based treatment and care as outlined in treatment guidelines and followed as usual at their local primary care center

INTERVENTIONS:
Behavioral: Person-centred care at distance through an eHealth platform — Person-centred care at distance through an eHealth platform, used by professionals, patients and relatives
  Arms: Person-centred care

SUMMARY:
The goal of the research project EAPER-P is to evaluate PCC person-centred care (PCC) in the form of a combined eHealth and telephone support for patents with chronic pain. A developed PCC eHealth platform, together with person-centred telephone conversations, will be used as a tool to identify patients´ resources to enhance coping and living with their illness by means of a dialog and partnership with staff and relatives. PCC in the form of a combined eHealth and telephone support will not replace, but instead be used as add on treatment to usual care (guideline directed care).

In addition, a process evaluation of the intervention will be performed in order to evaluate the mechanisms behind the intervention and evaluate which parts of the interventions the participants find useful.

DETAILED DESCRIPTION:
Previous research and collaboration between patients, relatives and professionals in the research program has clarified the need to develop a PCC accessible at home. Previous research has shown that eHealth support, where the users are not involved in the process, has a low impact and has highlighted several limitations with respect to patients' participation in the design process; its anchorage in the home and local environment and opportunities for communication rather than information. Therefore, this project has a participatory design that assumes that all users (patients, relatives and health care professionals) are involved in the study design, which facilitates implementation. An end-user perspective as a starting point increases the chances that users adapt a positive attitude towards the new system. PCC along the chain of health care showed a 4-fold chance of improved self-efficacy in combination with return to work or prior activity level after an event of acute coronary syndrome.

The aim of this project is to evaluate if PCC in the form of a combined eHealth and structured telephone support combined with an eHealth support available at home will improve return to work rates, reduced relapse, reduce costs and improved self-efficacy for patients with chronic pain.

This study is a randomized, open, parallel group intervention study where patients on sick leave for chronic pain are eligible. Patients will be randomized into either the control or the intervention arm 1:1. The control group will receive usual care. The intervention group will receive usual care plus PCC in the form of a combined eHealth and structured telephone support combined with an eHealth support. Randomization will be done through computer-generated lists and stored in sealed envelopes.

Patients listed in primary care with a confirmed diagnosis of chronic pain will be screened and sent an informing letter about the study from the chief at each center. Specially trained registered nurses (RNs) will then screen patients against study inclusion and exclusion criteria and by phone contact eligible patients and inform the patient about the aims of the study and ask if they are interested to participate. If the patient wants to participate, a consent form is sent to the patient and then returned to the RN. Written informed consent will then be obtained. Then the randomization procedure is performed which is stratified for age. The patient will be informed about the outcome by phone. Patients randomized to the intervention group will need a computer, smart phone or iPad with internet access to participate in the study. Patients randomized to usual care will be managed by regular evidence-based treatment and care as outlined in treatment guidelines and followed as usual at their local primary care center.

In PCC, the goals, capabilities and needs of each patient, will be the starting point. Self-care strategies will be reinforced and empowered. Patients in the intervention group will be contacted by a RN who has received special training in PCC communication for an initial person-centered dialogue by phone. The RN presents the eHealth platform and the RN invites the patient and activates their account where he/she can login via an individual user name.

During this phone conversation, the participants will also be invited to tell their story. Based on the patient narrative the patient´s goals, resources and needs are identified. The patient (sometimes maybe together with relatives) and the RN formulate a person-centered health plan. This plan is part of and will be up-loaded to the eHealth platform, which also contains individual notes and information about stress, depression and anxiety. The plan will be the point of departure for the forthcoming dialogue at distance via the eHealth platform that the patient and the RN will have during the study period (6 months).

The eHealth support contains headings that may inspire the patient to make notes on "a good day" respectively "a bad day" and register daily health related status. The health plan contain three parts; 1. "My goal is to feel or be able to do". 2. "To be able to reach my goal I will." 3."Support I need to reach my goal". In the communication during the study period between the RN and patient, the personal health plan is discussed and any needs of reformulating the goals may be discussed. The overall goal is to help the patient to identify their own capabilities/resources such as a strong will, social relations etc. and formulate goals that help them increase their self-efficacy and to cope with their condition in daily life.

At the end of each phone conversation, the participant and RN will agree on when and how they will be in contact next. I addition to these pre-agreed on phone conversations, the participants are free to contact the RNs via the eHealth platform or direct phone number.

On the eHealth platform, the participants can and formulate, comment, evaluate and develop the health plan, rate and follow their symptoms and keep a diary. Access to the eHealth platform will be password protected. The RN can see the patient´s account and make comments. The participants can invite other health care professionals, family and friend that they want to give access to the eHealth platform. The participants can add or delete these invitees when they want and they can limit the access for each invitee. The RNs follow the procedures closely. A monitor controls the protocol adherence. All case record forms, questionnaires and referrals will be constructed (for intervention and usual care groups).

Questionnaires on for example general self-efficacy, quality of life, anxiety and depression, symptom burden and daily functional level will be sent to all patients in both groups at inclusion and 3 months, 6 months, 1 year, 2 years and 5 years after randomization. In addition, data from registries, the platform and medical records will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years old.
* Living with chronic, non-malignant, pain with any of the following diagnoses: M25, M54, M79 and R52
* On sick leave (full or part time) from paid professional work.
* Willing to participate

Exclusion Criteria:

* Full time sick leave >24 months (part time sick leave >24 months can be included).
* Severe impairment (cognitive or other) that prevents patient from using the eHealth support
* No registered address
* Not willing to participate
* Any severe disease with an expected survival <12 months
* Ongoing documented diagnosis of alcohol or drug abuse
* Other severe disease that can interfere with follow-up or if the intervention is assessed as a burden
* Patient participating in another conflicting randomized study
* Patients not understanding spoken and written Swedish
* Patient not having access to a device with internet access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Composite score of changes | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  A patient is classified as improved, deteriorated or unchanged:
  A patient is classified as improved if:
  at 6 months reduced sick leave and increased General self-efficacy scale by ≥ 5 units
  A patient is classified as deteriorated if:
  at 6 months increased sick leave or (if on full-time sick leave at inclusion reduced general self-efficacy by ≥ 5 units)
  Those who have neither deteriorated nor improved are considered unchanged
  General Self-Efficacy Scale: Possible scores range from 10 (low self-efficacy, worst) to 40 (high self-efficacy).
  Composite score possible scores: deteriorated (worst), unchanged, improved (best).

SECONDARY OUTCOMES:
Sick leave | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Grade of sick leave Possible scores range from 0% (best) to 100% (worst)
General self-efficacy scale | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire General Self-Efficacy Scale: Possible scores range from 10 (low self-efficacy, worst) to 40 (high self-efficacy).
EuroQol- 5 Dimensions (EQ-5D) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire
  Possible scores on the different dimensions:
  Mobility I have no problems in walking about (best) I have some problems in walking about I am confined to bed (worst)
  Self-care I have no problems with self-care (best) I have some problems washing or dressing myself I am unable to wash or dress myself (worst)
  Usual activities (e.g. work, study, housework, family or leisure activities) I have no problems with performing my usual activities (best) I have some problems with performing my usual activities I am unable to perform my usual activities (worst)
  Pain/discomfort I have no pain or discomfort (best) I have moderate pain or discomfort I have extreme pain or discomfort (worst)
  Anxiety/depression I am not anxious or depressed (best) I am moderately anxious or depressed I am extremely anxious or depressed (worst)
  EQ-5D Visual Analog Scale (VAS) Possible range: 0 (the worst health you can imagine) to 100 (the best health you can imagine)
Hospital anxiety and depression scale (HADS) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire Total score possible range: 0 (best) to 42 (worst) Sub-scale depression possible range 0 (best) to 21 (worst) Sub-scale anxiety possible range 0 (best) to 21 (worst)
Number of health care visits (Health care utilization) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Health care utilization, data from registry where individual use of health care is recorded. Number of visits to health care. Ranges from 0 visits (best) and up. There is no maximum number of possible visits. More visits are worse.
Cost of health care utilized | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Health care utilization, data from registry where individual use of health care is recorded. Cost of health care visits ranges $0 (best) and up.There is no maximum cost of possible visits. Higher costs are worse.
Incremental cost-utility ratios | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Incremental cost-utility ratios
Tampa scale of kinesiophobia (TSK-SV) Possible score range from 17 (best) to 68 (worst) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire
Pain Disability Index (PDI) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire Possible score range from 0 (best) to 70 (worst)
Insomnia Severity Index (ISI) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire Possible score range from 0 (best) to 28 (worst)
Physical activity according to the Swedish National Board of Health and Welfare | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire Physical exercise possible range 0 (0 minutes of / week) to 6 (>120 minutes / week) Everyday physical activity possible range: 0 (0 minutes of / week) to 7 (>300 minutes / week)
Numeric Rating Scale for Pain (NRS Pain) | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire At rest possible score 0 (no pain) to 10 (worst possible pain) In motion possible score 0 (no pain) to 10 (worst possible pain)
The Being Taken Seriously Questionnaire | Baseline, 3 months, 6 months, 1 year, 2 years, 5 years.
  Questionnaire Possible score 6 (worst) to 48 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wallström, PhD, Principal Investigator — Göteborg University
Locations (1):
- Primary care, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No